CLINICAL TRIAL: NCT03092843
Title: Functional Capacity and Quality of Life Following SePtal Myectomy in patIents With Obstructive hypeRtrophIc cardiomyopaThy
Brief Title: Functional Capacity and Quality of Life Following Septal Myectomy in Patients With HCM
Acronym: SPIRIT-HCM
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Milind Desai, MD, The Cleveland Clinic
Other Study IDs: 17-176
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No functional capacity testing: 6 minute walk Quality of life Questionaire
- Functional Capacity Testing: 6 minute walk Quality of Life Questionnaire Metabolic stress test

SUMMARY:
Investigators aim to assess changes in exercise capacity and quality of life after septal myectomy in patient with hypertrophic cardiomyopathy.

DETAILED DESCRIPTION:
The objective of this study is to examine change in quality of life and functional capacity as respectively measured by, Quality of Life Questionnaires and six-minute walk test distance, following septal myectomy in patients with obstructive hypertrophic cardiomyopathy, as compared to prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo septal myectomy.
* Established diagnosis of obstructive HCM defined as:

LVH Thickness ≥15mm left ventricular outflow tract gradient ≥50mmHg

Exclusion Criteria:

* Prior septal myectomy or alcohol septal ablation
* Prior myocardial infarction
* Uncontrolled arrhythmias including ventricular tachycardia and atrial fibrillation
* Uncontrolled hypertension
* Angiographically documented coronary stenosis >50%, if available at time of screening
* Inability to provide informed consent
* Inability to walk without assistive devices
* Peripheral artery disease with claudication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-65 with an established diagnosis of obstructive hypertrophic cardiomyopathy and scheduled for septal Myectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life Change in Summary Score | 1 year post myectomy
  Mild improvement in Quality of Life summary score (increase in 5 points) as measured by Kansas City Cardiomyopathy Questionnaire -KCCQ

SECONDARY OUTCOMES:
Change in Quality of Life Change in Patient Reported Outcomes | 1 year post myectomy
  Quality of Life as measured by The Patient-Reported Outcomes Measurement Information System (PROMIS) Questionnaire
Change in Quality of Life Change in Duke's Activity Status Index (DASI) | 1 year post myectomy
  Quality of Life as measured by the Duke's Activity Status Index (DASI) Questionnaire
Change in functional capacity post myectomy | 1 year post myectomy
  Functional capacity will be measured by 6 minute walk

CONTACTS AND LOCATIONS:
Overall Officials: Milind Desai, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desai MY, Szpakowski N, Tower-Rader A, Bittel B, Fava A, Ospina S, Xu B, Thamilarasan M, Mentias A, Smedira NG, Popovic ZB. Echocardiographic Changes Following Surgical Myectomy in Severely Symptomatic Obstructive Hypertrophic Cardiomyopathy: Insights From the SPIRIT-HCM Study. J Am Heart Assoc. 2025 Jan 7;14(1):e037058. doi: 10.1161/JAHA.124.037058. Epub 2024 Dec 24. PMID 39719417
- [Derived] Tower-Rader A, Szpakowski N, Popovic ZB, Bittel B, Fava A, Ospina S, Xu B, Thamilarasan M, Mentias A, Smedira NG, Desai MY. Patient reported outcomes in obstructive hypertrophic cardiomyopathy undergoing myectomy: Results from SPIRIT-HCM study. Prog Cardiovasc Dis. 2023 Sep-Oct;80:66-73. doi: 10.1016/j.pcad.2023.06.001. Epub 2023 Jun 9. PMID 37302651